CLINICAL TRIAL: NCT00623025
Title: Double-blind, Cross-over, Randomized, Placebo-controlled, Multi-center Study to Investigate the Effect of Creon®25 000 on the Coefficient of Fat Absorption of HIV-infected Patients
Brief Title: Creon in HIV Patients With Steatorrhea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinued prematurely due to low enrollment
Sponsor: Abbott (Industry)
Responsible Party: Suntje Sander, Director Clinical Development, Abbott
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S245.3.125; 2007-005433-11 (EudraCT Number); 00623025 (Other: NCT/NIH)
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Steatorrhea
Keywords: HIV; Steatorrhea
MeSH Terms: conditions — Steatorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Creon 25000
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Creon 25000 — 6 to 9 capsules Creon 25000 per day
  Arms: 1
Drug: Placebo — 6 to 9 capsules placebo per day
  Arms: 2

SUMMARY:
The study investigates the effect of pancreatic enzymes on steatorrhea in HIV patients.

ELIGIBILITY:
Inclusion Criteria HIV positive patients with clinically stable disease (Karnofsky Performance Status > 40);

* Steatocrit > 2 %;
* Females of child-bearing potential must have a negative pregnancy test during prestudy or the subject must be surgically sterile or be at least 1 year postmenopausal as judged by the investigator;
* Women of child-bearing potential must be using a medically acceptable method of birth control throughout the study

Exclusion Criteria

* Known allergy to pancreatin or any history of abnormal drug reaction;
* Known diagnosis of pancreatic exocrine insufficiency due to e.g. chronic pancreatitis or cystic fibrosis or pancreatectomy;
* Intake of an experimental drug within four weeks prior to entry into the study;
* Alcohol abuse within the last six months;
* Suspected non-compliance or non-cooperation;
* Any other lack of fitness, in the investigator's opinion, to participate in or to complete the study;
* Patients with a stool fat excretion <= 7 g/day according to van de Kamer during the run-in period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Coefficient of fat absorption (CFA) | After 2 weeks

SECONDARY OUTCOMES:
Stool fat excretion | After 2 weeks
Normalization (yes, no) of stool fat excretion, i.e. < 7 g/day | After 2 weeks
Response (yes, no) with respect to stool fat excretion, i.e. improvement in stool fat excretion as compared to baseline | After 2 weeks
Stool weight | After 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suntje Sander, PhD, Study Director — Abbott
Locations (2):
- Romania (2):
  - Site Reference ID/Investigator# 59364, Bucharest
  - Site Reference ID/Investigator# 59363, Craiova